CLINICAL TRIAL: NCT00693264
Title: The Hemodynamic and Electrocardiographic Effects of Hoodia Gordonii in Healthy Volunteers
Brief Title: Effects of Hoodia on Blood Pressure and Heart Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Nickole Henyan/Assistant Professor of Pharmacy Practice, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2008-0005
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Healthy
Keywords: Human Volunteers; Hoodia; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will take 1- 750 mg capsule of Hoodia gordonii and have the primary and secondary outcomes measured over an 8 hour visit.
  Interventions: Dietary Supplement: Hoodia Gordonii
- 2 (Placebo Comparator): Participants will take a placebo capsule and have the primary and secondary outcome measures taken over an 8 hour study day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hoodia Gordonii — 750 mg capsule will be taken one time
  Other Names: Desert Burn
  Arms: 1
Dietary Supplement: Placebo — Placebo capsule to be taken one time
  Arms: 2

SUMMARY:
The purpose of the study is to learn about an herbal product called Hoodia gordonii. We want to know if Hoodia gordonii affects blood pressure, heart rate (pulse), heart pressures, and the heart's electrical conduction system. To participate in this study you must be a healthy volunteer with no known medical problems.

DETAILED DESCRIPTION:
If you decide to join this research study you will come in for two visits one week apart. Each visit will last 8 hours (you will not be required to stay in the exam room for the entire day). During the first visit you will be assigned, by chance, like the flip of a coin, to get either Hoodia gordonii or placebo. A placebo is a pill that looks like the herbal supplement but does not have any active ingredients in it. During the second visit you will get either Hoodia or placebo, whichever you did not get during the first visit. Neither you nor your study doctor will know ahead of time if you will get Hoodia or placebo during the first visit.

If you choose to participate in this study you have the following tests performed.

A. Electrocardiogram (ECG): this is a test that measures the electrical activity in the heart. This test involves placing 10 stickers on the chest and stomach and will last about 1 minute.

B. Blood Pressure: this is a test that involves placing a cuff on your arm and inflating it. Blood pressure cuffs might make you feel uncomfortable when they inflate, but it is not painful. The cuff will be placed on your arm for approximately 3 minutes.

C. Hemodynamics: these are tests that measure the pressures in the heart. This test involves placing 4 stickers (2 on your neck and 2 on your stomach) and is done while lying down. This test will last about 3 minutes and will be done at the same time as the blood pressure test.

Each test (A through C) will be performed a total of 10 times (5 times each study visit). Women of child bearing age will be required to take a urine pregnancy test. Pregnant women are not eligible to participate in this study. An outline of a study day is provided below.

1. Arrive at the exam room. ECG, Blood Pressure, and Hemodynamics are measured (for example, 8:00am).
2. Take the study pill (for example, 8:15am).
3. Return to exam room 1 hour after taking the study pill to have ECG, Blood Pressure, and hemodynamics measured (for example, 9:15am).
4. Return to the exam room 3 hours after taking the study pill to have ECG, Blood Pressure, and hemodynamics measured (for example, 11:15am).
5. Return to the exam room 5 hours after taking the study pill to have ECG, Blood Pressure, and hemodynamics measured (for example, 1:15pm).
6. Return to the exam room 8 hours after taking the study pill to have ECG, Blood Pressure, and hemodynamics measured (for example, 4:15pm).

Return to exam room 1 week later and repeat the day outlined above. Your participation in this study will last 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at least 18 years of age and in general good health expressing interest in participating in the study will be evaluated for inclusion.

Exclusion Criteria:

* baseline heart rate less than 50 beats/minute or greater than 100 beats/minute
* heart rhythm other than normal sinus
* history of atrial or ventricular arrhythmia
* family history of premature sudden cardiac death
* left ventricular hypertrophy
* atherosclerosis
* hypertension
* palpitations
* T-wave abnormality
* baseline corrected QT(QTc) interval greater than 440 milliseconds (ms)
* thyroid disease
* type 1 or 2 diabetes mellitus
* recurrent headaches
* depression
* any psychiatric condition or neurological disorder
* history of alcohol or drug abuse
* renal or hepatic dysfunction
* concurrent use of potentially interacting drugs (anticoagulants, MAO inhibitors, CYP 3A impacted drugs (substrate, inducer, or inhibitor) over the counter medications containing pseudoephedrine, caffeine containing products, or any dietary supplements)
* subject unwillingness to sign informed consent
* Pregnant or lactating females will also be also excluded from participation with urine dipstick tests used to confirm lack of pregnancy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the electrocardiographic effect, primarily the effect on the PR and RR intervals of H. gordonii in healthy individuals. | Baseline, 1, 3, 5 and 8 hours after taking study drug

SECONDARY OUTCOMES:
Evaluate other electrocardiographic effects, specifically effects on the QTc, QRS, and Tpe intervals of H. gordonii in healthy individuals. | Baseline, 1, 3, 5, and 8 hours after taking study drug
Evaluate the impact of H. gordonii on the following hemodynamic parameters: Blood Pressure, Cardiac Output, Systemic Vascular Resistance, and Thoracic Fluid Content. | Baseline, 1, 3, 5, and 8 hours after taking study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Nickole N Henyan, PharmD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States